CLINICAL TRIAL: NCT01931436
Title: A Single-site, Single-dose and Multiple-dose Study to Evaluate the Pharmacokinetics of the Main Components of Qing'E Pill (a Chinese Medicine Formula) Into the Blood in Chinese Menopausal Women
Brief Title: Pharmacokinetics Study of Qing'E Pill
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: QE-2458-2
Record Dates: First submitted 2013-08-08; First posted 2013-08-29 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Menopause
Keywords: Menopause, pharmacokinetic
MeSH Terms: interventions — Qing'e pill

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Qing'E pill (Experimental): Administered twice a day, and each 9 g
  Interventions: Drug: Qing'E pill

INTERVENTIONS:
Drug: Qing'E pill — Qing'E pill is composed of eucommia, psoralen, walnuts and garlic.

SUMMARY:
This study will investigate the pharmacokinetics of single and multiple doses of Qing'E pills in Chinese menopause volunteers. The main components of Qing'E pill into the blood such as psoralen and Isopsoralen will be detected.

ELIGIBILITY:
Inclusion Criteria:

1. Women age between 40 to 60 Years, Suffering from irregular menstrual cycle or amenorrhea of 3-11 months.
2. Moderate to severe hot flashes (associated with sweating)≥5 times /24 hours.
3. The score of Kupperman index is not less than 15.
4. Patients unused estrogen tablets or progesterone injection in 6 months.
5. Patients must discontinue other therapies in the treatment of menopausal syndrome for more than 3 months.
6. Get subjects informed consent process should comply with GCP requirements.

Exclusion Criteria:

1. There is no clinical significance abnormal in physical and laboratory examination.
2. Bilateral oophorectomy, endometrial lesions, uterine polyps, abnormal vaginal bleeding, severe breast hyperplasia, with family history of breast cancer.
3. Patients with hypertension, primary hypotension and chronic anemia (Hb ≤ 90 g/L).
4. Patients with hyperthyroidism, coronary atheroma, diabetes, obesity (body mass index of more than 30 kg/m2), migraine, malignant tumors, thromboembolic disease, gastrointestinal diseases affect absorption or autoimmune diseases.
5. Patients with diseases of the cardiovascular, cerebrovascular, liver, kidney and hematopoietic system, or mentally ill.
6. People with allergies.
7. People taking other drugs within 14 days before the trail.
8. Patients are participating in other clinical trials within 3 months.
9. Pregnant Women.
10. Alcoholics or smokers (past or smoking).

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of the main components of Qing'E pill (Maximum plasma concentration (Cmax), Area under the plasma concentration curve (AUClast and AUC)) | Up to 48 hours postdose for each period
  To detect the main components of Qing'E pill into the blood such as psoralen and Isopsoralen.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China